CLINICAL TRIAL: NCT00788918
Title: Study of Cerebral Function in Patients With Chronic Hepatitis C Infection Before and After Pegylated Interferon Alfa-2a and Ribavirin Therapy
Brief Title: Study of Cerebral Function in Patients With Chronic Hepatitis C Infection (HCV/CNS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SKS-0078-HCVCNS; EudraCT 2007-005707-18
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis C, Chronic; Cognition Disorders; Fatigue Syndrome, Chronic; Major Depressive Disorder
Keywords: Chronic Hepatitis C; cognitive dysfunction; MRI; MR spectroscopy; interferon; ribavirin; sustained virologic response, major depressive disorder
MeSH Terms: conditions — Hepatitis C, Chronic; Cognition Disorders; Fatigue Syndrome, Chronic; Depressive Disorder, Major; Cognitive Dysfunction | interventions — Interferons; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Chronic hepatitis C treatment (Experimental): 30 Chronic HCV patients with pending antiviral treatment. A majority will have pending treatment with interferon and ribavirin, and the treated patients will be assessed 8-12 weeks after starting treatment for interferon-induced depression.
  Interventions: Drug: Interferon and ribavirin
- Healthy Controls (No Intervention): 50 age, sex and education matched controls (matched 1:1 to participants in the HCV patient groups (+/- treatment)
- Former HCV infected (No Intervention): 20 Subjects with prior HCV infection identified through positive HCV antibodies, but negative HCV RNA.
- Chronic HCV patient - no treatment (No Intervention): 20 chronic HCV patients without pending antiviral treatment.

INTERVENTIONS:
Drug: Interferon and ribavirin — Interferon 180 microgram weekly s.c. and ribavirin (800/100/1200 mg daily) p.o.
  Other Names: Pegasys (ATC Code: L03AB11) and Copegus (ATC Code: J05AB04)
  Arms: Chronic hepatitis C treatment

SUMMARY:
Patients with HCV infection often suffer from chronic fatigue, depression and reduced cognition, even before evolving severe liver fibrosis, liver cirrhosis and hepatic encephalopathy.

It is currently unclear to what extent the symptoms er due to a direct pathological effects of the virus itself, or due to pre-existing psychiatric disease. There is a complex relationship between prior or existing drug abuse, psychiatric disease and HCV infection, that makes it difficult to establish cause-effect relationships.

A biological mechanism has been suggested to contribute to development of cerebral dysfunction in the patients. According to the prevailing Trojan Horses hypothesis circulating lymphocytes cross the blood brain barrier carrying HCV to the central nervous system and virus is subsequently replicated in the macrophages and the microglia in brain as a separate compartment. As part of the immunological response to viral replication, neurodegenerative processes takes place with a harmful effect on the neural circuit and cerebral function. Identification of HCV RNA negative strand, a replication product, in brain tissue from HCV patients, as part of autopsy studies, supports the hypothesis. Moreover, HCV patients have also been observed with abnormal metabolic concentrations in the frontal white substance and the basal ganglia by MRI spectroscopy compared to control groups.

The overall study objective is to assess cerebral function with particular emphasis on cognitive functions in HCV patients (genotypes 1,2,3 and 4) by use of a neuropsychiatric test battery. Furthermore, the patients will be examined by MRI, including magnetization transfer, diffusion tensor and contrast perfusion, in order to perform measurements of cerebral volumetric and microstructure. Finally, HCV analysis, including viral sequences and cytokine profiles, in serum and cerebrospinal fluid will be carried out in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection with genotype 1, 2, 3 or 4.
* Age > 18 and <60
* Liver biopsy or fibroscan performed within last 5 years
* Signed informed consent form.

Exclusion Criteria:

* Liver biopsy showing liver pathology not due to HCV infection.
* Liver cirrhosis or severe liver fibrosis
* Former antiviral HCV treatment (for included HCV patients).
* HIV and/or Hepatitis B virus infection.
* Alcohol or drug abuse within the last 2 years.
* Neutropenia, anemia or thrombocytopenia.
* Clinical signs of non-compensated liver pathology.
* Moderate to severe cardiopulmonary disease (NYHA score 1 or above)
* Creatinine clearance < 80mL/min.
* Pregnancy.
* Ferromagnetic implants
* Significant somatic disease affecting the central nervous system (somatic/neurologic disease)
* Head trauma resulting in unconsciousness > 5min
* Schizophrenia or other psychotic disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Neuropsychological test results, cytokine profile and MRI findings | 8 weeks before starting IFN+RIB therapy
  Assessment performed before starting antiviral treatment in patients with chronic hepatitis C who awaits treatment. HCV patients without pending treatment will be tested in conjunction with their outpatient controls.

SECONDARY OUTCOMES:
Interferon-induced depression | 8-12 weeks after treatment inititation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leutscher, MD, PhD, Principal Investigator — Aarhus University Hospital, Dept. Infectious Diseases
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Skejby, Aarhus, Jylland, Denmark

REFERENCES:
- [Background] Perry W, Hilsabeck RC, Hassanein TI. Cognitive dysfunction in chronic hepatitis C: a review. Dig Dis Sci. 2008 Feb;53(2):307-21. doi: 10.1007/s10620-007-9896-z. Epub 2007 Aug 17. PMID 17703362
- [Background] Forton DM, Hamilton G, Allsop JM, Grover VP, Wesnes K, O'Sullivan C, Thomas HC, Taylor-Robinson SD. Cerebral immune activation in chronic hepatitis C infection: a magnetic resonance spectroscopy study. J Hepatol. 2008 Sep;49(3):316-22. doi: 10.1016/j.jhep.2008.03.022. Epub 2008 Apr 25. PMID 18538439
- [Background] McAndrews MP, Farcnik K, Carlen P, Damyanovich A, Mrkonjic M, Jones S, Heathcote EJ. Prevalence and significance of neurocognitive dysfunction in hepatitis C in the absence of correlated risk factors. Hepatology. 2005 Apr;41(4):801-8. doi: 10.1002/hep.20635. PMID 15793853
- [Background] Golden J, O'Dwyer AM, Conroy RM. Depression and anxiety in patients with hepatitis C: prevalence, detection rates and risk factors. Gen Hosp Psychiatry. 2005 Nov-Dec;27(6):431-8. doi: 10.1016/j.genhosppsych.2005.06.006. PMID 16271658
- [Background] Laskus T, Radkowski M, Adair DM, Wilkinson J, Scheck AC, Rakela J. Emerging evidence of hepatitis C virus neuroinvasion. AIDS. 2005 Oct;19 Suppl 3:S140-4. doi: 10.1097/01.aids.0000192083.41561.00. PMID 16251811
- See also: Center for Functionally Integrative Neuroscience, Aarhus University Hospital — http://www.cfin.au.dk/
- See also: Center for Psychiatric Research, Aarhus University Hospital — http://psykiatriskforskning.dk/